CLINICAL TRIAL: NCT02959307
Title: Transcranial Continuous and Pulse Near-Infrared Light in Depression: a Placebo-Controlled Study (ELATED-3).
Brief Title: Transcranial Laser Therapy, Continuous and Pulsed Light, for Major Depressive Disorder (ELATED-3)
Acronym: ELATED-3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: LiteCure LLC (Industry)
Responsible Party: Principal Investigator, Paolo Cassano, Assistant Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2016P001490
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Results first posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-08

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder; Major Depressive Episode
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transcranial Light Therapy (Experimental): Transcranial light therapy penetrates the skin and brain using light energy and, the light energy may activate under-stimulated brain regions.
  Interventions: Device: Transcranial Light Therapy
- Sham Transcranial Light Therapy (Sham Comparator): For the sham group, The transcranial light therapy device uses nonpenetrating light emitting diode light energy. The sham controls for which participants improve from the actual transcranial light therapy treatment and which participants improve during the study for reasons other than the therapy
  Interventions: Device: Transcranial Light Therapy; Device: Sham Transcranial Light Therapy

INTERVENTIONS:
Device: Transcranial Light Therapy — Transcranial light therapy penetrates the skin and brain using light energy; this makes transcranial light therapy noninvasive. Transcranial light therapy may activate under-stimulated brain regions.
  Other Names: Low Level Laser-Light Therapy, Photobiomodulation
Device: Sham Transcranial Light Therapy — The same device used for the actual transcranial light therapy is used as the sham device; The device, when set to sham, will mimic the actual transcranial light therapy; however, when set to sham the device does not emit skin and cranium penetrating light emitting diode light energy.
  Other Names: Placebo
  Arms: Sham Transcranial Light Therapy

SUMMARY:
Transcranial Light Therapy involves non-invasive and invisible beams of light that increase energy metabolism in the brain. Transcranial light therapy has been found to promote brain metabolism which may help people with depression. The research team proposes a novel approach to treating depression by using transcranial light therapy.

DETAILED DESCRIPTION:
During study visits a clinician applies transcranial light therapy to both sides of a participant's forehead for about 30 minutes. The study involves, 1 screening visit which may last up to the 3 hours, 24 transcranial light therapy treatment visits, and 1 post-treatment visit (26 total visits to the Massachusetts General Hospital).

If a participant qualifies for the study, we assign the participant by chance to receive either active transcranial light therapy or sham transcranial light therapy treatment. During sham transcranial light therapy visits, the transcranial light therapy device will not produce near infrared waves (e.g., light energy that cannot penetrate the skin and cranium). Participants have an equal chance of being assigned to the active transcranial light therapy or the sham transcranial light therapy when first randomized. Neither the participant, nor the clinician, nor any research staff will know which study group the participant belongs.

Participants are randomized a second time after 6-weeks in the study. If the participant were in the sham group the first 6-weeks, that participant may receive the active transcranial light therapy treatment after re-randomization. If the participant were already in the active transcranial light therapy group during the first 6-weeks the participant continues receiving the active treatment. All in all, participants have a 1 in 3 chance of receiving the active transcranial light therapy treatment at some point during the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant age at screening will be between (>=)18 and 70 years old (inclusive).
* Participant meets the criteria for major depressive disorder
* Participants informed consent obtained in writing
* Participant is available to participate in the study for at least 12 weeks

Exclusion Criteria:

* Significant skin conditions near the application site
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment
* Recent history of stroke
* The participant failed more than 2 adequate treatment with Federal Drug Administration approved antidepressants during current episode per antidepressant treatment response questionnaire criteria (less than 50% decrease in depressive symptomatology).
* Structured psychotherapy focused on treating the subject's depression (i.e. cognitive behavioral therapy or interpersonal therapy) is permitted if started at least 8 weeks prior to the screening visit.
* Substance dependence or abuse in the past 3 months.
* History of a psychotic disorder or psychotic episode (current psychotic episode per M.I.N.I neuro-psychiatric assessment).
* Bipolar affective disorder (per M.I.N.I neuro-psychiatric assessment).
* Unstable medical illness, defined as any medical illness which is not well-controlled with standard-of-care medications (e.g., insulin for diabetes mellitus, hydrochlorothiazide for hypertension).
* Active suicidal or homicidal ideation (both intention and plan are present), as determined by Columbia Suicide Severity Rating Scale
* Cognitive impairment (Montreal Cognitive Assessment <21)
* The participant has a significant skin condition (i.e., hemangioma, scleroderma, psoriasis, rash, open wound or tattoo) on the subject's scalp that is found to be in proximity to any of the procedure sites.
* The subject has an implant of any kind in the head (e.g. stent, clipped aneurysm, embolised arteriovenous malformation, implantable shunt - Hakim valve).
* Any use of light-activated drugs (photodynamic therapy) within 14 days prior to study enrollment (in US: Visudyne (verteporfin) - for age related macular degeneration; Aminolevulinic Acid- for actinic keratoses; Photofrin (porfimer sodium) - for esophageal cancer, non-small cell lung cancer; Levulan Kerastick (aminolevulinic acid hydrogen chloride) - for actinic keratosis; 5-aminolevulinic acid for non-melanoma skin cancer)
* Women of child-bearing potential must use a double-barrier method for birth control (e.g. condoms plus spermicide) if sexually active.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cassano, M.D., Principal Investigator — Depression Clinical and Research Program
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York

IPD SHARING:
Plan to Share IPD: Yes
Personally unidentifiable information will be sent to Dr. Anastasia Ivanova, a privately contracted biostatistician form Chapel Hill North Carolina, for analyses. All information sent to Dr. Ivanova uses acrostics in place of personally identifiable information.

REFERENCES:
- [Derived] Iosifescu DV, Norton RJ, Tural U, Mischoulon D, Collins K, McDonald E, De Taboada L, Foster S, Cusin C, Yeung A, Clain A, Schoenfeld D, Hamblin MR, Cassano P. Very Low-Level Transcranial Photobiomodulation for Major Depressive Disorder: The ELATED-3 Multicenter, Randomized, Sham-Controlled Trial. J Clin Psychiatry. 2022 Aug 8;83(5):21m14226. doi: 10.4088/JCP.21m14226. PMID 35950904

RESULTS

PARTICIPANT FLOW:
Period: Phase 1
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
Started | 18 | 31
Completed | 15 | 23
Not Completed | 3 | 8
Period: Phase 2
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
Started | 28 (This group is increased as those in sham were re-randomized to sham or NIR.) | 10 (This group is decreased as those in sham were re-randomized to sham or NIR.)
Completed | 26 | 10
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy | Total
Number analyzed (Participants) | 18 | 31 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.222 (15.509) | 42.806 (15.823) | 40.755 (16.137)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 4 | 10 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 15 | 25 | 40
  Unknown or Not Reported | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 13 | 27 | 40
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Age of Depressive Onset [Mean (Standard Deviation); unit: years] — Participants were asked when they first remembered onset of depressive symptoms. Some participants had trouble recollecting. Analysis was only performed on participants who had definitive age of onset.
  years | 17.294 (9.973) | 23.429 (16.089) | 21.111 (14.285)

OUTCOME MEASURES:

1. Primary Outcome: Quick Inventory of Depressive Symptomatology-Phase 1
Description: This is a brief (16-item) clinician-rated inventory of core depressive symptoms such as sleep, depressed mood, appetite, concentration, suicidal ideation, interest, energy, psychomotor retardation or agitation. Scores range from 0-27, higher scores indicating greater depression severity.
Time Frame: 6 weeks - Sequential-parallel comparison design
Population: Sham Group in Phase 1 accounts for all subjects Receiving Sham. Patients in Sham within the first phase would be re-randomized to either NIR or Sham after completion of the initial 6 weeks. 2 participants in Sham did not have scores collected, as such the Sham group for Phase 1 consists of 29 participants rather than the total 31.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
Number analyzed (Participants) | 18 | 29
score on a scale | 11.06 (3.78) | 11.24 (4.83)

2. Primary Outcome: Quick Inventory of Depressive Symptomatology(QIDS)-Phase 2
Description: as for outcome 1
Time Frame: 6 weeks - Sequential-parallel comparison design
Population: This group consists of all sham participants that did not respond to Sham in Phase 1 and were re-randomized into Phase 2. Therefore, of the 29 participants in Sham, 5 participants were responders, 4 were not re-randomized.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
Number analyzed (Participants) | 11 | 7
score on a scale | 10.45 (5.751) | 9.14 (5.551)

3. Secondary Outcome: Hamilton Depression Rating Scale - 17 Items(Phase 1)
Description: assessment of the patient's depressive symptoms, using a structured interview and defined anchor points. The Hamilton Depression Rating Scale aims to quantify the degree of depression in patients who already have a diagnosis of major depression. Score ranges from 0-52. Higher score indicates greater severity of depression.
Time Frame: 6 weeks - Sequential-parallel comparison design
Population: Patients in Sham within the first phase would be re-randomized to either NIR or Sham after completion of the initial 6 weeks. There were two participants in the Sham group who did not have scores for the primary analysis (QIDS), we decided to include them in the secondary analysis (HAMD) as they had scores.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
Number analyzed (Participants) | 18 | 31
score on a scale | 16.28 (5.345) | 15.81 (6.685)

4. Secondary Outcome: Hamilton Depression Rating Scale - 17 Items(Phase 2)
Description: as for outcome 3
Time Frame: 6 weeks - Sequential-parallel comparison design
Population: This group consists of all sham participants that did not respond to Sham in Phase 1 and were re-randomized into Phase 2. Therefore, of the 29 participants in Sham, 5 participants were responders, 4 were not re-randomized. 1 participant was not assessed with HAMD but was assessed with primary measure (QIDS), as such there are 10 in TLT group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
Number analyzed (Participants) | 10 | 7
score on a scale | 13.50 (6.151) | 14.14 (6.768)

ADVERSE EVENTS:
Time Frame: Timeframe of collection was during participation in the two phases of the study and follow up visit 1 week after completion. Therefore, the total timeframe of assessment is 13 weeks.
Description: Our participants flow differs for the following reasons: Per the SPCD design, subjects within the Sham group in Phase 1 are re-randomized in Phase 2 to receive either Sham or TLT treatment. Therefore, TLT group accounts for participants receiving TLT in the first phase as well as those re-randomized to TLT in their second phase. Participants in Sham account for all subjects randomized to sham in Phase 1, regardless of whether they were re-randomized to Sham or TLT in Phase 2.
Arm/Group | Transcranial Light Therapy | Sham Transcranial Light Therapy
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/31 | 1/31
Other Adverse Events (participants affected / at risk) | 12/31 | 17/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcranial Light Therapy (N=31) | Sham Transcranial Light Therapy (N=31)
Aborted Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1) — Aborted suicide attempt that triggered a hospitalization while participant was outside of lab.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Transcranial Light Therapy (N=31) | Sham Transcranial Light Therapy (N=31)
Headache (General disorders) | 9 | 7
Worsening of Pre-Existing Condition (General disorders) | 3 | 3
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Insomnia (Psychiatric disorders) | 5 | 4
Irritability With and Without Impulsivity (Psychiatric disorders) | 1 | 4
Panic Attack (Psychiatric disorders) | 1 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Pressure on Forehead/Head (General disorders) | 4 | 2

LIMITATIONS AND CAVEATS:
For the device utilized in this trial, very low light was applied. In addition, two nodes were obstructed by participants' hair, reducing light delivered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT02959307/Prot_000.pdf
  • Informed Consent Form (2017-03-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT02959307/ICF_001.pdf
  • Statistical Analysis Plan (2020-05-12): https://cdn.clinicaltrials.gov/large-docs/07/NCT02959307/SAP_002.pdf